CLINICAL TRIAL: NCT00058825
Title: Phase I/II Study of Allogeneic Stem Cell Transplantation for Patients With Hematologic Diseases Using Haploidentical Family Donors and Sub-Myeloablative Conditioning With Campath 1H
Brief Title: Stem Cell Transplant for Hematologic Diseases
Acronym: HIMSUM
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Slow accrual due to practice changes meant study would take too long to finish
Sponsor: Baylor College of Medicine (Other)
Collaborators: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, George Carrum, Principal Investigator, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8713-HIMSUM
Record Dates: First submitted 2003-04-11; First posted 2003-04-15 (Estimated); Results first posted 2015-10-22 (Estimated); Last update posted 2016-11-07 (Estimated); Status verified 2016-09

CONDITIONS: Hematologic Malignancies
Keywords: Campath; stem cell transplant
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Alemtuzumab; fludarabine; Stem Cell Transplantation; Whole-Body Irradiation; Tacrolimus; Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stem Cell Transplant (Experimental): Total body irradiation (TBI); Fludarabine and Campath 1H; FK506 or Cyclosporine; Stem Cell Transplant; G-CSF.
  Interventions: Biological: Campath 1H; Drug: Fludarabine; Procedure: Stem Cell Transplant; Radiation: Total Body Irradiation (TBI); Drug: FK506 (Tacrolimus) or Cyclosporine

INTERVENTIONS:
Biological: Campath 1H — Day -5 to Day -2: Campath 1H dose schedule as per institutional SOP.
Drug: Fludarabine — Day -5 to Day -2: Fludarabine 30 mg/m2.
Procedure: Stem Cell Transplant — Day 0: Donor stem cells infused.
Radiation: Total Body Irradiation (TBI) — Day -6: Total body irradiation of 600 cGy as two doses without blocks at a rate of less than or equal to 10 cGy/minute.
Drug: FK506 (Tacrolimus) or Cyclosporine — Day -2: FK506 or Cyclosporine as medically indicated to prevent GvHD.

SUMMARY:
Patients are being asked to participate in this study because they have a cancer in their blood, Fanconi's Anemia, or have been unsuccessfully treated for bone marrow failure such as Aplastic Anemia or Paroxysmal Nocturnal Hemoglobinuria. Any of these conditions could benefit from an allogeneic stem cell transplant using a donor that is related to the patient.

Stem cells are created in the bone marrow. They grow into different types of blood cells that the patient needs, including red blood cells, white blood cells, and platelets. In a transplant, the patient's own stem cells are killed and then replaced by stem cells from the donor.

Usually, patients are given very strong doses of chemotherapy prior to receiving a stem cell transplant. However, because of the patient's condition, they have a high risk of experiencing life-threatening treatment-related side-effects. Recently, some doctors have begun to use chemotherapy that does not cause as many side-effects before patients receive a transplant.

This research study adds CAMPATH 1H to a low-dose chemotherapy regimen, followed by an allogeneic stem cell transplantation. We want to see whether adding CAMPATH 1H to the transplant medications helps in treating the disease. We also want to see whether there are fewer life-threatening side-effects from the treatment. CAMPATH 1H is a drug that is still being studied. CAMPATH 1H stays active in the body for a long time after patients receive it, which means it may work longer at preventing graft-versus-host-disease (GvHD) symptoms.

DETAILED DESCRIPTION:
Before treatment begins, stem cells will be collected from the donor's blood or bone marrow. The stem cells will be collected and frozen before we start to give the patient chemotherapy.

After admission to the hospital, patients will receive total body irradiation (very strong x-rays that kill cells in the bone marrow), Fludarabine and Campath 1H prior to the stem cell transplant (infusion of the donor's stem cells).

Starting 7 days after the transplant, the patient will be given G-CSF by subcutaneous injection, until a blood test shows that numbers of granulocytes (a type of white blood cell) in the blood are more than 1,000/uL. This is to help increase blood cell counts.

After transplantation, the patient will undergo several evaluations at different times. These are standard evaluations and tests performed for any patient who has received a stem cell transplant, as part of routine clinical monitoring.

We will also be looking at the patient's immune function (how the body protects itself to prevent and fight infections and diseases). To do this, blood tests will be performed at regular intervals (every 3 to 6 months) for 2 years.

Depending on how well the donor stem cells work in the body after the transplant, the patient may receive one or more Donor Leukocyte Infusions (DLI). This is when leukocytes (a type of white blood cell) collected from the same donor that provided the stem cells are given to the patient through a central line into a vein.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Diagnosis of myelodysplastic disorders; Fanconi's Anemia; Acute Myelogenous Leukemia (including secondary); Acute Lymphoblastic Leukemia; Multiple Myeloma; Plasma Cell Dyscrasia; lymphoproliferative disorders (Non-Hodgkin Lymphoma, Hairy Cell Leukemia, Chronic Lymphocytic Leukemia, and Hodgkin's Disease). Diagnosis of myelodysplastic disorders which is not good risk by IPSS: Fanconi's Anemia; Acute Myelogenous Leukemia (1st or subsequent relapse, or 2nd or subsequent CR, or refractory disease); Acute Lymphoblastic Leukemia in 2nd or subsequent remission or relapse or refractory disease; Philadelphia Chromosome-positive Chronic Myelogenous Leukemia (failed STI and interferon); Multiple Myeloma (Stage II or III); Lymphoma; Chronic Lymphocytic Leukemia (primary refractory or recurrent disease); Hodgkin's Disease (after relapse); Hemophagocytic Lymphohistiocytosis (failed chemotherapy and/or anti-viral therapy); bone marrow failure such as Aplastic Anemia and Paroxysmal Nocturnal Hemoglobinuria; PNH (failed prior therapies).
2. Conditions that increase treatment related mortality: (need one or more to be eligible): Age > / = 50 years; EF of less than 45%; DLCO less than 50% or FEVI 50-75% of predicted value; Diabetes Mellitus; Renal Insufficiency (but creatinine clearance not less than 25 mL/min); Prior recent history of systemic fungal infection; 3rd or greater remission of AML or ALL; Significant Grade III or IV neurologic or hepatic toxicity from previous treatment; More than 1 year from diagnosis (CML or Myeloma patients ONLY); Multiple types of treatment regimens (equal to or more than 3); Significant Grade III or IV neurologic or hepatic toxicity from previous treatment; Prior autologous or allogeneic stem cell transplantation.
3. Haploidentical family member donor. This protocol is open to patients who lack a 5/6 or 6/6 HLA antigen-matched donor. Due to the increased risk of GvHD, patients with Fanconi Anemia and a 5/6 HLA match will also be eligible.

   For this protocol, the "best" donor will be defined as a first-degree haploidentical family member who matches at the greatest number of MHC loci. Matching will be determined by Class I and Class II DNA typing. The donor should be sufficiently healthy as to not be at increased risk from the stem cell mobilization procedure. Should more than one "equally" MHC-incompatible donor be identified, other selection criteria will include: age and size of donor, CMV status, and sex. The Principal Investigator will make final decisions.
4. Available healthy donor without any contraindications for donation.
5. Patient and/or legal representative and/or legal guardian able to understand and sign consent.
6. Age between birth and 70 years.
7. Women of child-bearing potential must have a negative pregnancy test.

EXCLUSION CRITERIA:

1. Pregnant, lactating or unwilling to use contraception.
2. HIV-positive patient.
3. Uncontrolled intercurrent infection.
4. Untreated blast crisis for CML.
5. Uncontrolled high-grade lymphoproliferative disease / lymphoma.
6. Unstable angina and uncompensated congestive heart failure (Zubrod of 3 or greater).
7. Severe chronic pulmonary disease requiring oxygen (Zubrod of 3 or greater).
8. Hemodialysis dependent.
9. Active hepatitis or cirrhosis with total bilirubin, SGOT, and SGPT greater than 3X upper limit of normal.
10. Unstable cerebral vascular disease and recent hemorrhagic stroke (less than 6 months).
11. Active CNS disease from hematological disorder.

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2000-08; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Carrum, MD, Principal Investigator — Baylor College of Medicine; The Methodist Hospital
Locations (2):
- United States (2):
  - Texas Children's Hospital, Houston, Texas
  - The Methodist Hospital, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Stem Cell Transplant
Started | 27
Completed | 5
Not Completed | 22
Not completed — Relapse | 9
Not completed — Progressive Disease | 5
Not completed — Graft Failure | 5
Not completed — Death | 3

BASELINE CHARACTERISTICS:
Arm/Group | Stem Cell Transplant
Number analyzed (Participants) | 27
Age, Continuous [Median (Full Range); unit: years] | 15 [2 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Transplant Related Mortality (TRM)
Description: Percentage of patients with transplant related mortality
Time Frame: 100 days
Measure: Number (97.5% Confidence Interval); unit: percentage of participants
Arm/Group | Stem Cell Transplant
Number analyzed (Participants) | 27
percentage of participants | 0 [0 to 12.8]

2. Secondary Outcome: Time in Days to ANC Engraftment
Description: Engraftment was defined as the day of absolute neutrophil counts (ANC) exceeded 0.5 X 10^9/L on the first of 3 days.
Time Frame: 30 days
Measure: Median (Full Range); unit: days
Arm/Group | Stem Cell Transplant
Number analyzed (Participants) | 27
days | 12 [6 to 21]

3. Secondary Outcome: Donor Chimerism Engraftment of Greater Than 50%
Description: Number of patients that engrafted who showed a chimerism (donor cells) of greater than 50% in the first 30 days
Time Frame: 30 days
Population: Patients engrafted
Measure: Number; unit: participants
Arm/Group | Stem Cell Transplant
Number analyzed (Participants) | 22
participants
  Yes | 20
  No | 2

4. Secondary Outcome: Acute Graft Versus Host Disease
Description: Number of patients with Acute Graft Versus Host Disease within 100 days post-transplant
Time Frame: 100 days
Measure: Number; unit: participants
Arm/Group | Stem Cell Transplant
Number analyzed (Participants) | 27
participants
  Grade 0 | 26
  Grade I | 0
  Grade II | 0
  Grade III | 1
  Grade IV | 0

5. Secondary Outcome: Chronic Graft Versus Host Disease
Description: Number of patients with Chronic Graft Versus Host Disease within 1 year post-transplant
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Stem Cell Transplant
Number analyzed (Participants) | 27
participants
  Yes | 1
  No | 26

6. Secondary Outcome: 2-year Relapse-free Survival
Description: Relapse-free survival (RFS) was calculated from the time of transplant to the date of relapse, death, or last follow-up, whichever occurred first. Survival data were analyzed by Kaplan-Meier method.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stem Cell Transplant
Number analyzed (Participants) | 27
percentage of participants | 25.9 [11.5 to 43.1]

7. Secondary Outcome: 2-year Overall Survival
Description: Overall survival (OS) was calculated from the time of transplant to death from any cause or censored at last follow-up. Survival data were analyzed by Kaplan-Meier method.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stem Cell Transplant
Number analyzed (Participants) | 27
percentage of participants | 33.3 [16.8 to 50.9]

8. Secondary Outcome: Number of Patients Who Engrafted With the Isolex/CLINIMACs System
Description: Engraftment was defined as the day of absolute neutrophil counts (ANC) exceeded 0.5 X 10^9/L on the first of 3 days.
Time Frame: 30 days
Measure: Number; unit: participants
Groups:
- Isolex: The Isolex system was used for cell selection.
- CLINIMACs: The CLINIMACS CD34 Reagent system was used for cell selection.
Arm/Group | Isolex | CLINIMACs
Number analyzed (Participants) | 19 | 8
participants | 15 | 7

9. Secondary Outcome: Median Time to Engraftment With the Isolex/CLINIMACs System
Description: Engraftment was defined as the day of absolute neutrophil counts (ANC) exceeded 0.5 X 10^9/L on the first of 3 days.
Time Frame: 30 days
Measure: Median (Full Range); unit: days
Arm/Group | Isolex | CLINIMACs
Number analyzed (Participants) | 19 | 8
days | 12 [6 to 21] | 12 [9 to 17]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected until 30 days after autologous transplants and until 100 days after allogeneic transplants.
Arm/Group | Stem Cell Transplant
Serious Adverse Events (participants affected / at risk) | 4/27
Other Adverse Events (participants affected / at risk) | 19/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stem Cell Transplant (N=27)
Failure to engraft (Blood and lymphatic system disorders) | 1 (1)
Infection (documented clinically or microbiologically) with grade 3 or 4 neutropenia (Infections and infestations) | 1 (1)
Infection without neutropenia (Infections and infestations) | 2 (4)
Hypokalemia (Metabolism and nutrition disorders) | 1 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stem Cell Transplant (N=27)
Failure to engraft (Blood and lymphatic system disorders) | 4 (4)
Transfusion: Platelets (Blood and lymphatic system disorders) | 7 (16)
Anorexia (Gastrointestinal disorders) | 7 (7)
Nausea (Gastrointestinal disorders) | 3 (7)
Vomiting (Gastrointestinal disorders) | 2 (5)
GGT (Gamma-Glutamyl transpeptidase) (Hepatobiliary disorders) | 3 (5)
SGPT (ALT) (serum glutamic pyruvic transaminase) (Hepatobiliary disorders) | 2 (4)
Catheter-related infection (Infections and infestations) | 2 (3)
Febrile Neutropenia (Infections and infestations) | 3 (3)
Infection (documented clinically or microbiologically) with grade 3 or 4 neutropenia (Infections and infestations) | 8 (11)
Infection without neutropenia (Infections and infestations) | 5 (12)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (3)
Hypokalemia (Metabolism and nutrition disorders) | 3 (5)
Abdominal Pain or Cramping (General disorders) | 2 (2)
Bone Pain (General disorders) | 3 (3)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes